CLINICAL TRIAL: NCT03707847
Title: Single-arm, Multi-center Clinical Study of Crizotinib Combined With Etoposide Capsule Followed by Auto-HSCT for Relapsed and Refractory Anaplastic Lymphoma Kinase (ALK)-Positive Anaplastic Large Cell Lymphoma (ALCL)
Brief Title: Crizotinib Combined With Etoposide Capsule Followed by Auto-HSCT for Relapsed and Refractory ALK+ ALCL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20180821
Record Dates: First submitted 2018-09-23; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: ALK-Positive Anaplastic Large Cell Lymphoma
Keywords: crizotinib; etoposide; autologous hematopoietic stem cell transplantation; ORR; OS; PFS; adverse events
MeSH Terms: interventions — Crizotinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Crizotinib + etoposide capsule+Auto-HSCT (Experimental): Crizotinib and etoposide capsule followed by autologous hematopoietic stem cell transplantation.
  Crizotinib: 250mg, bis in die （BID）, PO.
  Etoposide capsule:50mg, quaque die （QD）, PO, d1-10，21days for one cycle.
  Patients will receive the treatment of crizotinib and etoposide capsule, and those who have achieved CR（complete response）or VGPR（very good partial response）will undergo the Auto-HSCT.
  Interventions: Drug: Crizotinib; Drug: Etoposide Capsule; Procedure: Auto-HSCT

INTERVENTIONS:
Drug: Crizotinib — 250mg, BID, PO
Drug: Etoposide Capsule — 50mg, QD, PO, d1-10，21days for one cycle
Procedure: Auto-HSCT — Auto-HSCT will be performed with patients who have achieved CR or VGPR.

SUMMARY:
To observe the safety, tolerability and clinical effects of crizotinib combined with etoposide capsule followed by autologous hematopoietic stem cell transplantation (Auto-HSCT) for patients with relapsed and refractory ALK-positive Anaplastic Large Cell Lymphoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, one-arm, multicenter clinical trial, aimed to evaluate the safety, tolerability, and efficacy of crizotinib combined with etoposide followed by autologous hematopoietic stem cell transplantation for relapsed and refractory ALK-positive ALCL. A total of 20 patients are planned to be enrolled into the study. Patients with diagnosis of relapsed and refractory ALK-positive ALCL will be treated with crizotinib plus etoposide capsules followed by autologous hematopoietic stem cell transplantation. The primary end points are objective responder rate (ORR) and progression free survival(PFS) and the secondary end points include overall survival(OS) , and adverse events.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* age:14-65 years;Eastern Cooperative Oncology Group (ECOG)score≤3;expected survival≥3 months
* patients with ALK-positive Anaplastic Large Cell Lymphoma diagnosed by immuno-histochemistry (IHC) or fluorescence in situ hybridization (FISH);
* Refractory or relapse after at least 4 cycles of CHOP（cyclophosphamide, hydroxydaunomycin, Oncovin, and prednisone）regimen
* acceptable hematological indicators, no chemotherapy contraindications;
* total bilirubin ≤ 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 2.5 x upper age limit (ULN), if the abnormal laboratory parameters are considered to be caused by lymphoma, patients Eligible conditions should be adjusted to be incorporated into the group;
* At least one measurable lesion by CT or PET-CT（Positron Emission Tomography-Computed Tomography）;
* exclude other major diseases, normal heart and lung function;
* Female patients of childbearing age are negative for pregnancy test;
* Cooperate with follow-up;
* There are no other related treatments including traditional Chinese medicine, immunotherapy, and biologic therapy (except for the treatment of anti-bone metastases and other symptoms);
* Signing informed consent *: Pathological histology must be consulted by a pathologist at a provincial hospital.

Exclusion Criteria:

* rejecting providing blood preparation;
* allergic to drug in this study and with metabolic block;
* rejecting adopting reliable contraceptive method in pregnancy or lactation period;
* uncontrolled internal medicine disease(including uncontrolled diabetes,severe incompetence cardiac,lung,liver and pancreas）；
* with severe infection;
* with primary or secondary central nervous system tumor invasion;
* with immunotherapy or radiotherapy contraindication;
* ever suffered with malignant tumor;
* having peripheral nervous system disorder or dysphrenia;
* with no legal capacity,medical or ethical reasons affecting research proceeding;
* participating other clinical trials simultaneously;
* adopting other anti-tumor medicine excluding this research;
* Patients with immunodeficiency, such as primary immunodeficiency syndrome or organ transplant recipients
* Human immunodeficiency virus (HIV)-positive patients
* the researchers considering it inappropriate to participate in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  Objective Responder Rate
PFS | up to 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
OS | up to 24 months
  Overall Survival
adverse events | up to 24 months
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China